CLINICAL TRIAL: NCT04229004
Title: Precision Promise Platform Trial for Metastatic Pancreatic Cancer
Brief Title: A Multi-center Trial to Evaluate Multiple Regimens in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pancreatic Cancer Action Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PanCAN_Precision Promise
Record Dates: First submitted 2019-12-19; First posted 2020-01-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Gemcitabine combined with nab-paclitaxel (Active Comparator): Arm is closed to recruitment.
  The following are recommended parameters for infusion timing and sequence, although institutional variation in the administration of the regimen are permitted as long as drug dosing and modification guidelines are followed.
  Interventions: Drug: Gemcitabine combined with nab-paclitaxel
- mFOLFIRINOX (Active Comparator): Arm is closed to recruitment.
  Oxaliplatin 85 mg/m2, Leucovorin 400 mg/m2, Irinotecan 150 mg/m2, 5-Fluorouracil 2400 mg/m2 46-48 hour infusion
  Interventions: Drug: Dose -mFOLFIRINOX
- pamrevlumab (FibroGen) (Experimental): Arm is closed to recruitment.
  Experimental: Pamrevlumab in combination with gemcitabine/nab-paclitaxel.
  Participants enrolled to this treatment arm will receive treatment with pamrevlumab in combination with gemcitabine and nab-paclitaxel.
  Gemcitabine and nab-paclitaxel are FDA approved therapies for metastatic pancreatic cancer and will be supplied or obtained according to local clinical study agreements and in accordance with local guidelines.
  Interventions: Drug: Dose - Pamrevlumab combined with gemcitabine and nab-paclitaxel
- Canakinumab and Spartalizumab (Experimental): Arm is closed to recruitment.
  Canakinumab and Spartalizumab in Combination with Nab-Paclitaxel and Gemcitabine.
  Participants enrolled to this treatment arm will receive treatment with Canakinumab and Spartalizumab in combination with nab-paclitaxel and gemcitabine.
  Interventions: Drug: Dose- Canakinumab and Spartalizumab combined with nab-paclitaxel and gemcitabine
- Experimental: SM-88 (Experimental): Arm is closed to recruitment.
  460 mg (2 capsules) twice daily of a 28-day cycle along with the administration of methoxsalen, phenytoin and sirolimus.
  All four agents (SM-88, methoxsalen, phenytoin, and sirolimus) should be dosed with approximately 240 mL (8 fl. oz.) of water in the morning. All four agents should be taken together consistently. SM-88 used with MPS should ideally be taken approximately 1 hour before or 2 hours after a meal.
  Interventions: Drug: Drug: Dose -SM-88

INTERVENTIONS:
Drug: Gemcitabine combined with nab-paclitaxel — Arm is closed to recruitment.
  Nab-paclitaxel is infused over 30-40 min on days 1, 8, 15 of each 28-day cycle. Gemcitabine is infused over 30 min, immediately after completion of nab-paclitaxel infusion, on days 1, 8, 15 of each 28-day cycle.
  If one of the chemotherapy medications is held, the other study medications may be given.
  Doses should be re-adjusted if the participant's weight changes by +/- >10%. If the participant's weight changes by <10%, no adjustment is necessary unless the site has a standard procedure to adjust doses based upon current weight according to institutional guidelines.
  Arms: Gemcitabine combined with nab-paclitaxel
Drug: Dose -mFOLFIRINOX — Arm is closed to recruitment.
  The following are recommended parameters for infusion timing and sequence, although institutional variation in the administration of the regimen are permitted, as long as drug dosing and modification guidelines are followed. Oxaliplatin and leucovorin are administered concurrently over 30-120 minutes, followed by irinotecan over 30-90 minutes, followed by the infusion of 5-flurouracil. If one of the chemotherapy medications is held, the other study medications may be given. Doses should be re-adjusted if the participant's weight changes by +/- >10%. If the participant's weight changes by <10%, no adjustment is necessary unless the site has a standard procedure to adjust doses based upon current weight according to institutional guidelines.
  Arms: mFOLFIRINOX
Drug: Dose - Pamrevlumab combined with gemcitabine and nab-paclitaxel — Arm is closed to recruitment.
  Pamrevlumab 35mg/kg IV - Cycle 1 (Day 1, 8, 15 of the 28 day cycle) and Cycle 2 and Onward (Day 1 and 15)
  Nab-paclitaxel 125mg/m2 IV - Day 1, 8, 15 for every 28 day cycle
  Gemcitabine 1000mg/m2 IV - Day 1, 8, 15 for every 28 day cycle
  Arms: pamrevlumab (FibroGen)
Drug: Dose- Canakinumab and Spartalizumab combined with nab-paclitaxel and gemcitabine — Arm is closed to recruitment.
  Canakinumab 250mg SC- Day 1 of every 28 day cycle
  Spartalizumab 400 mg IV - Day 1 of every 28 day cycle
  Nab-paclitaxel 125mg/m2 IV - Day 1, 8, 15 of every 28 day cycle
  Gemcitabine 1000mg/m2 IV - Day 1, 8, 15 of every 28 day cycle
  Arms: Canakinumab and Spartalizumab
Drug: Drug: Dose -SM-88 — Arm is closed to recruitment.
  460 mg (2 capsules) twice daily of a 28-day cycle along with the administration of methoxsalen, phenytoin and sirolimus.
  Arms: Experimental: SM-88

SUMMARY:
Precision Promise is a multi-center, seamless Phase 2/3 platform trial designed to evaluate multiple regimens in metastatic pancreatic cancer.

Primary Objectives

* To compare each investigational arm versus standard of care (SOC) for superiority in overall survival in first and/or second line metastatic ductal adenocarcinoma (metastatic pancreatic cancer) participants and determine which, if any, participants benefit from each investigational arm.

Secondary Objectives

* To determine short and long-term safety signals of each investigational arm in metastatic pancreatic cancer participants vs. SOC.
* To determine progression-free survival (PFS) for each investigational arm vs. SOC.
* To determine rates of overall response, CR, and PR; duration of overall response, CR or PR (whichever occurs first).
* To determine rates of clinical benefit; duration of clinical benefit.

DETAILED DESCRIPTION:
Precision Promise is a multi-center, seamless Phase 2/3 platform trial designed to evaluate multiple regimens in metastatic pancreatic cancer. The goal of the platform is to find effective therapies for pancreatic cancer. The platform will test multiple investigational drugs and combinations compared to standard of care therapy in first and second line metastatic participants. Bayesian response-adaptive randomization will be used to assign participants to arms based on their performance in subtypes of the disease. The primary endpoint is overall survival.

ELIGIBILITY:
Inclusion Criteria

A participant will be eligible to participate in Precision Promise if all the below inclusion criteria are met:

* Age ≥ 18 years
* Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma (PDAC) and eligible for treatment in the first line or second line settings.
* Acceptable histologies include adenosquamous carcinoma, mucinous adenocarcinoma, hepatoid carcinoma, medullary carcinoma, signet ring cell carcinoma, undifferentiated carcinoma, and undifferentiated carcinoma with osteoclast-like-cells, and adenocarcinoma. Pancreatic neuroendocrine tumors (PNET) are excluded.
* Radiographically measurable disease by computed tomography (CT) scan or magnetic resonance imaging (MRI) as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Imaging results must be obtained within the 28-day window, prior to randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ function (lab results must be obtained within the 28-day window prior to randomization)

  * Absolute neutrophil count ≥ 1500/mm3
  * Hemoglobin ≥ the lower limit of normal (LLN) or 9g/dL
  * Platelets ≥ 100,000/mm3
  * Serum creatinine ≤ 1.0 x upper limit normal (ULN), or calculated creatinine clearance ≥ 50 mL/min (Cockcroft Gault)
  * Albumin ≥ 3.0 g/dL
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x ULN (up to ≤ 5 x ULN in presence of liver metastasis).
  * Total bilirubin ≤ 1.5 x ULN
  * INR ≤ 1.5 x ULN (up to ≤ 2 x ULN for participants on anticoagulation therapy).
* Participants must be willing to provide protocol-mandated tissue and blood samples for diagnostic and research purposes as a condition of enrollment into the trial.
* Able to swallow pills, capsules or tablets.
* Able to adhere to study visit schedule and other protocol requirements.
* Participants of childbearing potential [defined as a person assigned as female at birth who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)] must:

  * Have a negative serum or urine pregnancy test (β-human chorionic gonadotropin [β-hCG]) as verified by the study doctor within 14 days prior to randomization.
  * Commit to complete abstinence from sexual contact with persons assigned as male at birth or agree to use medical doctor-approved contraception without interruption while participating in the study, during dose interruptions and for at least 6 months following last dose of study treatment.
* Participants assigned as males at birth must practice complete abstinence or agree to use a condom (even if he has undergone a successful vasectomy) during sexual contact with persons of childbearing potential while participating in the study, during dose interruptions and for at least 6 months following last dose of study treatment.
* known HIV-infected participants on effective anti-retroviral therapy are eligible if the most recent viral load test performed within six months of screening (based on medical chart review) is negative. If this is not the case, an HIV viral load test should be performed at screening and be negative (i.e., undetectable).
* Known HBV-infected participants are eligible if the most recent viral load test performed within six months of screening (based on medical chart review) is negative. If this is not the case, an HBV viral load test should be performed at screening and be negative (i.e., undetectable).
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with known HCV infection who are currently on treatment are eligible if the most recent viral load test performed within six months of screening (based on medical chart review) is negative. If this is not the case, an HCV viral load test should be performed at screening and be negative (i.e., undetectable).
* Participants with a history of brain metastases are eligible provided they show evidence of stable lesions (and no new lesions) with no evidence of tumor progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. In addition, any neurological symptoms that developed either as a result of the brain metastases or their treatment, must have returned to baseline or resolved. Any steroids administered as part of this therapy must be completed > 7 days prior to the first dose of trial therapy.
* No known leptomeningeal disease.
* Participants with a prior or concurrent malignancy whose natural history does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible. Participants receiving any active therapy for a concurrent secondary malignancy are excluded.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using New York Heart Association Functional Classification. To be eligible for this trial, participants should be Class 2 or better. Class 2 is defined as slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest.
* Understands the nature of the study and has agreed to participate by voluntarily signing the IRB approved informed consent.

Exclusion Criteria

A participant will not be eligible to participate in Precision Promise if any of the following criteria are met:

* Received any anti-cancer systemic therapy within 21 days (or 5 half-lives, whichever is shorter,) prior to randomization.
* Has had major surgery within 14 days prior to enrollment.
* History of known allergy or hypersensitivity to any of the study treatments or any of their excipients or contraindication to any of the study treatments as outlined in the local prescribing information (e.g., United States Prescribing Information [USPI]).
* Pre-existing peripheral neuropathy > Grade 1, as defined by CTCAE V 4.03.
* Known active tuberculosis infection.
* Serious, non-healing wound, ulcer, or bone fracture.
* The inability to swallow pills, capsules or tablets.
* Receiving any active therapy for concurrent secondary malignancy. Participants with a prior or concurrent malignancy whose natural history and/or management does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible.
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, and pulmonary hypersensitivity pneumonitis.
* QTc > 450 msec if male and QTc > 470 msec if female.
* Uncontrolled or severe cardiac disease (history of unstable angina, myocardial infarction, coronary stenting, or bypass surgery within the prior 6 months), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia [including atrial flutter/fibrillation].
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using New York Heart Association Functional Classification. Participants worse than Class 2 are excluded. Class 2 is defined as slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest.
* Active, uncontrolled infections (bacterial, viral, or fungal infection(s)) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment (i.e., Participants must be afebrile for > 48 hours off antibiotics).
* Active, known or suspected autoimmune disease, including systemic lupus erythematosus, Hashimotos thyroiditis, scleroderma, polyarteritis nodosa or autoimmune hepatitis.

  o Participants with type I diabetes mellitus, hypothyroidism requiring only hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are eligible to participate.
* Receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the Investigator, increase the risk of serious neutropenic complications. Participants receiving replacement therapy of 10 mg of prednisone (or the equivalent hydrocortisone dose) per day are eligible.
* Receipt of live vaccines within 30 days prior to the first dose of study treatment or while on active treatment within the trial. (examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are permitted. However, intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not permitted).COVID-19 vaccines are permitted.
* Any significant medical condition, laboratory abnormality or psychiatric illness that would limit the participant's ability to comply with study requirements.
* Participants that discontinued previous treatment for pancreatic adenocarcinoma due to a treatment-related ≥ Grade 3 toxicity.

  o For toxicity ≤ Grade 3, AE(s) must resolve to Grade 1 or baseline in order to be considered eligible for this trial.
* Participants that have received allogenic bone marrow or solid organ transplants are excluded.
* Participants that are pregnant, planning on becoming pregnant, or are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 0 weeks
  Overall survival (OS) is defined from the time of initiation of treatment until death due to any cause. Participants still alive at the time of an analysis will be considered censored at their date of last contact.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From initiation of therapy to clinically determined disease progression or death due to any cause, whichever came first, assessed up to 24 months.
  PFS will be presented with probability that the hazard ratio is less than 1.0 as well as the corresponding Kaplan-Meier curves and the log-rank test for the comparison with controls.
Performance Status | From screening through study completion, an average of 2 years.
  Changes in Performance Status will be evaluated using the Eastern Cooperative Oncology Group (ECOG) Performance Status, where the highest value is 0 (patient is fully active) and the lowest value is 5 (patient is deceased).
Overall Response Rate (ORR) | From initiation of treatment to clinically determined tumor size reduction for a minimum of 4 weeks
  ORR is defined as the portion of subjects on an arm with a tumor size reduction of at least 30%.
Duration of Overall Response Rate (ORR) | From date of first occurrence of a documented objective response to date of clinically determined disease progression or death due to any cause, whichever came first, assessed up to 24 months.
  Duration of ORR is defined as the time from the date of response to the date of clinically determined disease progression or death due to any cause.
Duration of Clinical Benefit | From screening through last dose of therapy, assessed up to 24 months.
  Duration of Clinical Benefit will be evaluated using a composite of measures including patient reported outcomes (PROs), supportive care regimens, and disease status.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan - Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center (MCCC), Rochester, Minnesota
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - New York University Langone Medical Center - Perlmutter Cancer Center, New York, New York
  - Evelyn H. Lauder Breast Center - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Physicians - Solid Tumor/Gastrointestinal Oncology, New York, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
  - Virginia Mason Hospital & Seattle Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rayego-Mateos S, Morgado-Pascual JL, Lavoz C, Rodrigues-Diez RR, Marquez-Exposito L, Tejera-Munoz A, Tejedor-Santamaria L, Rubio-Soto I, Marchant V, Ruiz-Ortega M. CCN2 Binds to Tubular Epithelial Cells in the Kidney. Biomolecules. 2022 Feb 3;12(2):252. doi: 10.3390/biom12020252. PMID 35204752